CLINICAL TRIAL: NCT00027430
Title: TheraDerm Administration in Women With Hypopituitarism
Brief Title: Androgen Replacement Therapy in Women With Hypopituitarism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: FD-R-1981-01; FD-R-001981-01
Record Dates: First submitted 2001-12-05; First posted 2001-12-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-11

CONDITIONS: Hypopituitarism
MeSH Terms: conditions — Hypopituitarism

INTERVENTIONS:
Drug: TheraDerm

SUMMARY:
This is a study to determine whether testosterone replacement with TheraDerm can improve bone density, mood, sex drive, thinking, and distribution of body fat and muscle mass in women with hypopituitarism.

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups to receive testosterone replacement therapy or placebo. Group 1 will receive 2 testosterone patches and estrogen pills for 12 months. Group 2 will receive 2 placebo patches and estrogen pills for 12 months. Changes in bone density, bone metabolism markers, body composition, libido, and quality of life will be compared in the women receiving testosterone replacement therapy with that of the women receiving placebo.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Hypogonadism and/or hypoadrenalism of central origin
* Testosterone or free testosterone level below the median for age-matched normal controls
* Prior estrogen preparation for at least 6 months

Exclusion criteria:

* Any disease known to affect bone metabolism, including untreated hypothyroidism or hyperthyroidism
* Change in thyroid hormone dose in the last 3 months
* Untreated Cushing's syndrome
* Renal failure
* Alcoholism
* Anorexia nervosa
* Prior use of medication known to affect bone metabolism (e.g., supraphysiologic doses of glucocorticoids, phenytoin, bisphosphonates, or calcitonin) within the past 3 months
* Pregnant or nursing
* Uncontrolled hypertension
* ALT greater than 3 times upper limit of normal
* Serum creatinine greater than 2 times the upper limit of normal
* Any contraindication to estrogen therapy, including history of breast cancer or undiagnosed uterine bleeding
* Concurrent growth hormone replacement therapy, if patient has been receiving it for less than 2 years

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-09; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lin E, McCabe E, Newton-Cheh C, Bloch K, Buys E, Wang T, Miller KK. Effects of transdermal testosterone on natriuretic peptide levels in women: a randomized placebo-controlled pilot study. Fertil Steril. 2012 Feb;97(2):489-93. doi: 10.1016/j.fertnstert.2011.11.001. Epub 2011 Dec 2. PMID 22137497